CLINICAL TRIAL: NCT03257943
Title: A Multi-Center, Double-Blind, Randomized, Placebo Controlled, Parallel-group Study, Comparing Ivermectin Lotion, 0.5% in the Treatment of Subjects With Active Infestation With Head Lice and Their Ova
Brief Title: A Bioequivalence Study, Comparing Two Formulations of Ivermectin Lotion, 0.5%
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IVRL 1604
Record Dates: First submitted 2017-05-03; First posted 2017-08-22 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Lice; Head Lice
MeSH Terms: conditions — Lice Infestations | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ivermectin Lotion, 0.5% (Experimental): One 10 minute application, under at-home use conditions
  Interventions: Drug: Ivermectin Lotion, 0.5%
- SKLICE (ivermectin) Lotion, 0.5% (Active Comparator): One 10 minute application, under at-home use conditions
  Interventions: Drug: SKLICE (ivermectin) Lotion, 0.5%
- Vehicle of the Test product (Placebo Comparator): One 10 minute application, under at-home use conditions
  Interventions: Drug: Vehicle of the Test product

INTERVENTIONS:
Drug: Ivermectin Lotion, 0.5% — Ivermectin Lotion, 0.5% (Taro Pharmaceuticals Inc.)
  Other Names: ivermectin
  Arms: Ivermectin Lotion, 0.5%
Drug: SKLICE (ivermectin) Lotion, 0.5% — SKLICE (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)
  Other Names: ivermectin
  Arms: SKLICE (ivermectin) Lotion, 0.5%
Drug: Vehicle of the Test product — Vehicle for Ivermectin Lotion, 0.5% (Taro Pharmaceuticals Inc.)
  Other Names: placebo
  Arms: Vehicle of the Test product

SUMMARY:
A Multi-Center, Double-Blind, Randomized, Placebo controlled, Parallel-group study, comparing Ivermectin Lotion, 0.5%

DETAILED DESCRIPTION:
A Multi-Center, Double-Blind, Randomized, Placebo controlled, Parallel-group study, comparing Ivermectin Lotion, 0.5% to Sklice (Ivermectin) Lotion, 0.5% and both active treatment to a placebo control in the treatment of subjects with active infestation with head lice and their Ova

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age or older must have provided IRB-approved written informed consent and sign a HIPAA authorization.
* Subjects must be willing and able to understand and comply with the requirements of the protocol, including attendance at the required study visits.

Exclusion Criteria:

* Subjects with a history of hypersensitivity or allergy to or any component of the study product.
* Subject with history of irritation or sensitivity to pediculicides or hair care products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-06-27 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Demonstration of Bioequivalence in proportion of index subjects who are lice free | Day 15 (14 days after application of study treatment)
  Demonstration of Bioequivalence in proportion of index subjects who are lice free

CONTACTS AND LOCATIONS:
Overall Officials: Catawba Research, Study Chair — http://catawbaresearch.com/contact/
Locations (1):
- Taro Pharmaceuticals USA Inc., Hawthorne, New York, United States

IPD SHARING:
Plan to Share IPD: No